CLINICAL TRIAL: NCT05106374
Title: FITNESS: Calculating Risk of Chemotherapy Toxicity in Older Adults
Brief Title: Risk of Chemotherapy Toxicity in Older Patients With Blood Cancer or Non-small Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Ashley Rosko, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-18055; NCI-2020-01239 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Mental Status and Dementia Tests; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire, assessment, biospecimen): Patients complete questionnaires over 30-40 minutes about daily activity and feelings, complete thinking and walking tests over 10 minutes, and undergo collection of blood samples before the first dose of chemotherapy and 90, 180, and 365 days after first dose of chemotherapy. Patients with non-small lung cancer also undergo collection of stool sample.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
Procedure: Cognitive Assessment — Complete thinking test
Other: Physical Performance Testing — Complete walking test
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial evaluates the risk of chemotherapy toxicity in older patients with blood cancer or non-small cell lung cancer. The purpose of this study is to describe a patient's wellness before and after chemotherapy treatment. This may help researchers better understand patient's ability to tolerate treatment and in the future devise the best treatment for a patient based on their "fitness."

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To validate the accuracy and predictive ability of the Cancer and Aging Research Group (CARG) Chemo-Toxicity calculator in untreated patients with hematologic malignancy and non-small cell lung cancer, as well as relapsed patients with a hematologic malignancy intended to begin chimeric antigen receptor (CAR) T cell therapy.

Ia. Determine if the CARG Chemo-Toxicity calculator predicts grade 3-5 toxicity in older adult patients with hematologic malignancy undergoing treatment.

Ib. Determine if CARG Geriatric Assessment (GA) metrics predict grade 3-5 toxicity in older adults with hematologic malignancy undergoing treatment.

Ic. Identify the association between frailty metrics and relative dose intensity in older adults with hematologic malignancy.

Id. To evaluate feasibility of CARG GA and functional assessment implementation in older adults with non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To determine the relationship of frailty metrics (CARG chemo-toxicity calculator and geriatric assessment metrics) with health related quality of life (HRQL) over time.

II. To identify the relationship of frailty metrics (chemo-toxicity calculator and GA metrics) with physical function as measured by the short physical performance battery (SPPB).

III. To determine the association of molecular markers of aging (OSU_Senescence, Hovarth epigenetic clock/deoxyribonucleic acid [DNA]ge, inflammatory cytokines, changes in peripheral blood T lymphocyte subsets) with risk of chemotherapy toxicity using the Chemo-Toxicity calculator and other prognostic factors (e.g. age, disease, stage, body composition by imaging).

IV. In the NSCLC cohort we will determine the association between treatment efficacy and toxicity with changes in the stool microbiome.

OUTLINE:

Patients complete questionnaires over 30-40 minutes about daily activity and feelings, complete thinking and walking tests over 10 minutes, and undergo collection of blood samples before the first dose of chemotherapy and 90, 180, and 365 days after first dose of chemotherapy. Patients with non-small lung cancer also undergo collection of stool sample.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Untreated for a hematologic malignancy or NSCLC malignancy with intention to receive treatment (i.e., chemotherapy, immunotherapy, targeted agents, bone marrow transplant, or other) at the Ohio State University; or patients with a relapsed hematologic malignancy intended to begin CAR T cell therapy
* Ability to understand and willingness to sign an informed consent document (or indicate approval or disapproval by another means)

Exclusion Criteria:

* Prisoners are excluded from participation
* Any medical condition including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a hematologic malignancy and are either untreated or relapsed and newly diagnosed with NSCLC who intend to receive treatment at the Ohio State University
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognostic ability of the CARG chemotoxicity calculator in patients newly diagnosed with hematologic malignancy | 365 days after first dose of chemotherapy
Predictive ability of the Cancer and Aging Research Group (CARG) Chemo-Toxicity calculator | 365 days after first dose of chemotherapy
Predictive ability of Chemo-Toxicity calculator to predict grade 3-5 toxicity | 365 days after first dose of chemotherapy
  Will fit a Cox regression model for time to toxicity (grades 3-5) containing the baseline chemo-toxicity risk score as the only predictor. The overall ability of the model to distinguish grade 3-5 from grade 1-2 toxicity will be evaluated using Harrell's C-statistic, which can be viewed as a generalization of the area under the curve measurement for receiver operator characteristics (ROC's) curves based on binary outcome data. A 95% confidence interval will be constructed for the C-statistic and if the lower bound is greater than 0.5 (expected value if the risk score is not predictive of toxicity) we will conclude that risk score is significantly able to distinguish between toxicity grades.
Predictive ability of Geriatric Assessment (GA) metrics to predict grade 3-5 toxicity | 365 days after first dose of chemotherapy
  Will fit a Cox regression model for time to toxicity (grades 3-5) containing the baseline chemo-toxicity risk score as the only predictor. The overall ability of the model to distinguish grade 3-5 from grade 1-2 toxicity will be evaluated using Harrell's C-statistic, which can be viewed as a generalization of the area under the curve measurement for ROC's curves based on binary outcome data. A 95% confidence interval will be constructed for the C-statistic and if the lower bound is greater than 0.5 (expected value if the risk score is not predictive of toxicity) we will conclude that risk score is significantly able to distinguish between toxicity grades.
Association between frailty metrics and relative dose intensity (RDI) | 365 days after first dose of chemotherapy
  Will explore the relationship of RDI and MAX2 (reduced and prescribed) with clinical and biologic factors of frailty. RDI (>= 85% versus [vs.] < 85%) will be treated as a continuous and dichotomous variable. The distribution of RDI and MAX2 will be examined graphically and transformed to normality as appropriate. Linear regression for continuous RDI and logistic regression for dichotomized RDI will be used to understand the relationship with RDI and independent variables (e.g. GA scores, age, short physical performance battery [SPPB] etc.) Stepwise regression will be used to identify significant clinical and biologic factors (e.g. OSU_Senescence) that are independently associated with continuous or dichotomized RDI.

SECONDARY OUTCOMES:
Relationship of frailty metrics with health related quality of life over time | 365 days after first dose of chemotherapy
  Linear mixed models will be used in the analyses. Each model will include effects of each prognostic variable of interest, time (baseline vs. end of treatment), and time-by-prognostic variable interactions to determine if the associations between the prognostic variables and the outcome differs at baseline and end of treatment. An unstructured covariance matrix will be used to model the relationship between outcome measurements from the same patient.
Relationship of frailty metrics with physical function | 365 days after first dose of chemotherapy
  Linear mixed models will be used in the analyses. Each model will include effects of each prognostic variable of interest, time (baseline vs. end of treatment), and time-by-prognostic variable interactions to determine if the associations between the prognostic variables and the outcome differs at baseline and end of treatment. An unstructured covariance matrix will be used to model the relationship between outcome measurements from the same patient.
Molecular markers of aging with risk of chemotherapy toxicity using the Chemo-Toxicity calculator | 365 days after first dose of chemotherapy
  Will determine the association of molecular markers of aging with risk of chemotherapy toxicity using the Chemo-Toxicity calculator and other prognostic factors (e.g. age, disease, stage, body composition by imaging). Linear mixed models will be used in the analyses. Each model will include effects of each prognostic variable of interest, time (baseline vs. end of treatment), and time-by-prognostic variable interactions to determine if the associations between the prognostic variables and the outcome differs at baseline and end of treatment. An unstructured covariance matrix will be used to model the relationship between outcome measurements from the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley E Rosko, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu